CLINICAL TRIAL: NCT00766662
Title: Intermittent Preventive Treatment in Infant in Mali
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bamako (Other)
Collaborators: UNICEF (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 06-55
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-09

CONDITIONS: Malaria
Keywords: Malaria; Intermittent Preventive Treatment; EPI vaccine coverage; Resistance of P. falciparum to Sulfadoxine- Pyrimethamine
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sulfadoxine pyrimethamine

SUMMARY:
Studies have shown that Intermittent preventive treatment in infants (IPTi) with Sulfadoxine-pyrimethamine (SP)reduced the incidence of clinical malaria and anemia without modifying infants' serological response to EPI vaccines. Thus IPTi was seen as a potential public health tool of great benefit to the children of Africa and a logical addition to the Immunization Plus package. The objectives of this operational researcher were

* to develop an implementation model for IPTi in the health care system in Mali
* to assess its impact on the EPI vaccines and other health interventions coverage
* and on molecular makers of resistance to SP

DETAILED DESCRIPTION:
The study was implemented in districts of the region of Koulikoro; the district of Koulikoro and the district of Kolokani. The whole district of Koulikoro was covered by the intervention while in Kolokani, the 22 health areas (sub districts) were randomized in 1:1 ratio with the intervention in 11 health areas and the other 11 serving as control for the assessment of the impact of IPTi implementation on EPI vaccines and other health interventions coverage as well as its impact on the resistance to SP. The implementation consisted of administration of ½ tablet of Sulfadoxine -Pyrimethamine with EPI vaccines (DTP2, DTP3 and Measles vaccine) from December 2006 to December 2007.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Kolokani, Mali
* Age less than 24 months

Exclusion Criteria:

* Not Resident of Kolokani
* Age of 24 months or above

Max Age: 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
EPI vaccines and other health interventions coverage | 1 year
Molecular makers of resistance of P. falciparum to Sulfaxodine- pyrimethamine | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alassane Dicko, MD, Principal Investigator — Faculty of Medicine, Pharmacy and Dentistry; University of Bamako; Ogobara K Doumbo, MD, Study Director — Faculty of Medicine, Pharmacy and Dentistry; University of Bamako
Locations (1):
- Malaria Research & Training Center; Faculty of Medicine, Pharmacy and Dentistry, University of Bamako, Bamako, Mali

REFERENCES:
- [Derived] Dicko A, Konare M, Traore D, Testa J, Salamon R, Doumbo O, Rogier C. The implementation of malaria intermittent preventive trialtreatment with sulphadoxine-pyrimethamine in infants reduced all-cause mortality in the district of Kolokani, Mali: results from a cluster randomized control. Malar J. 2012 Mar 16;11:73. doi: 10.1186/1475-2875-11-73. PMID 22423611
- [Derived] Dicko A, Toure SO, Traore M, Sagara I, Toure OB, Sissoko MS, Diallo AT, Rogier C, Salomon R, de Sousa A, Doumbo OK. Increase in EPI vaccines coverage after implementation of intermittent preventive treatment of malaria in infant with Sulfadoxine -pyrimethamine in the district of Kolokani, Mali: results from a cluster randomized control trial. BMC Public Health. 2011 Jul 18;11:573. doi: 10.1186/1471-2458-11-573. PMID 21767403